CLINICAL TRIAL: NCT04915391
Title: Restenosis in Coronary Stents And Cutaneous HEaling: Identification of Biochemical Markers and Potential Therapeutic Targets
Brief Title: Restenosis in Coronary Stents And Cutaneous HEaLing
Acronym: RACHEL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Responsible Party: Sponsor
Other Study IDs: RACHEL
Record Dates: First submitted 2021-03-16; First posted 2021-06-07 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-07

CONDITIONS: Coronary Restenosis; Coronary Stent Occlusion; Skin Scarring; Keloid
Keywords: Restenosis; Keloid; Hypertrophic skin scarring
MeSH Terms: conditions — Coronary Restenosis; Cicatrix; Keloid | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Two skin biopsies of the shoulder and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of controls: Control group of 40 patients with ≥1 bare metal stent which in a posterior catheterization performed by clinical follow-up had no restenosis
  Interventions: Diagnostic Test: Skin biopsy and blood sample for inflammation markers, RNA and proteins
- Group of cases: Group of cases with 20 patients with ≥1 bare metal stent and 20 patients with ≥1 drug eluting stent which had restenosis in a posterior catheterization performed by clinical follow-up.
  Interventions: Diagnostic Test: Skin biopsy and blood sample for inflammation markers, RNA and proteins

INTERVENTIONS:
Diagnostic Test: Skin biopsy and blood sample for inflammation markers, RNA and proteins — A skin biopsy will be performed at the baseline visit from which primary cell cultures of fibroblasts and keratinocytes will be obtained. Four to six weeks later a second biopsy on the scar will be performed and analyzed anatomically and pathologically. In addition, at the initial visit, blood samples will be drawn for analysis of inflammation markers, RNA and proteins.

SUMMARY:
Case control study of patients with and without restenosis to demonstrate the link between in-stent restenosis and an excessive skin healing. Patients will undergo skin biopsy and blood sample tests to search for a relationship between both processes and for the identification of biomarkers and therapeutic targets.

DETAILED DESCRIPTION:
Restenosis represents an excessive response to the coronary stent. On the other hand, skin healing with keloid formation is also an excessive repair response. There is evidence that both processes may be related because they share mechanisms mediated by inflammatory response. The purpose is to demonstrate the correlation between them for the identification of biomarkers and therapeutic targets.

The project is a case-control study with 2 groups of patients: a control group of 40 patients with ≥1 bare metal stent which in a posterior catheterization performed by clinical follow-up had no restenosis and a group of 20 patients with ≥1 bare metal stent and 20 patients with ≥1 drug eluting stent which had restenosis in a posterior catheterization also performed by clinical follow-up.

A skin biopsy will be performed at the baseline visit from which primary cell cultures of fibroblasts and keratinocytes will be obtained. Four to six weeks later a second biopsy on the scar will be performed and analyzed anatomically and pathologically. In addition, at the initial visit, blood samples will be drawn for analysis of inflammation markers, RNA and proteins. Studies can be performed at 3 levels:

1. The similarities and differences in cutaneous healing of patients with and without restenosis will be studied in the samples from the second biopsy.
2. With the cell culture from the first biopsy, the investigators will analyze the response of cutaneous cells to antiproliferative drugs and the potential advantage of vitamin D in inhibiting restenosis.
3. With the blood samples the investigators will analyze inflammatory factors, RNA and proteins that can predict these processes and that, in addition, can become potential therapeutic targets which might reduce the rate of restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous coronary stent implantation and a posterior catheterization performed > 8 months after the index procedure due to clinical follow-up (those ones with bare metal stents without restenosis will be included in the group of controls and those with restenosis will be included in the group of cases, 20 with bare metal and 20 with drug eluting stents).
* Age 18-75 years.

Exclusion Criteria:

* Patients on chronic anti-inflammatory treatment, including corticosteroids.
* Patients with previous or current history of malignancy or any other disease mediated by inflammation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bare metal stents without restenosis will be included in the group of controls and those with restenosis will be included in the group of cases, 20 with bare metal and 20 with drug eluting stents).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Link between in-stent restenosis and excessive skin healing | Through study completion, an average of 1 year
  Percentage of patients in case and control groups with hypertrophic pattern of skin healing after the first biopsy

SECONDARY OUTCOMES:
Response of skin cells to antiproliferative drugs | Through study completion, an average of 1 year
  Comparison of the proliferation rate of primary skin fibroblasts, from patients of the different groups, undergoing treatment with an antiproliferative drug. The continuous variable will be the percentage of living cells at the end of the treatment with respect to the initial cells, and mean values in the groups will be statistically compared.
Circulating microRNA profile | Through study completion, an average of 1 year
  Determination of the profile and levels of circulating microRNAs in patients from the different groups. Plasma samples from some individuals in each group will be analyzed using a microarray. To assess the level of circulating microRNAs in all patients, real-time reverse transcription-polymerase chain reaction will be used. Mean values in the groups will be statistically compared.
Blood levels of immune cell subsets related to vascular repair and endothelial damage, including antiogenic T-cells, immunosenescent T-cells, monocyte subsets and low-density granulocytes. | Through study completion, an average of 1 year
  These populations will be measured in samples of peripheral blood or isolated mononuclear cells by flow cytometry according to the expression of their surface markers

CONTACTS AND LOCATIONS:
Overall Officials: Iñigo Lozano, MD, PHD, Principal Investigator — Hospital Cabuenes
Locations (1):
- Department of Cardiology, Hospital Cabueñes, Gijón, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Komatsu R, Ueda M, Naruko T, Kojima A, Becker AE. Neointimal tissue response at sites of coronary stenting in humans: macroscopic, histological, and immunohistochemical analyses. Circulation. 1998 Jul 21;98(3):224-33. doi: 10.1161/01.cir.98.3.224. PMID 9697822
- [Result] Ozdol C, Turhan S, Tulunay C, Altin AT, Atmaca Y, Candemir B, Erol C. Association between proliferative scars and in-stent restenosis. J Cutan Med Surg. 2007 Nov-Dec;11(6):206-10. doi: 10.2310/7750.2007.00039. PMID 18042333
- [Result] Kornowski R, Hong MK, Tio FO, Bramwell O, Wu H, Leon MB. In-stent restenosis: contributions of inflammatory responses and arterial injury to neointimal hyperplasia. J Am Coll Cardiol. 1998 Jan;31(1):224-30. doi: 10.1016/s0735-1097(97)00450-6. PMID 9426044
- [Result] Albinsson S, Suarez Y, Skoura A, Offermanns S, Miano JM, Sessa WC. MicroRNAs are necessary for vascular smooth muscle growth, differentiation, and function. Arterioscler Thromb Vasc Biol. 2010 Jun;30(6):1118-26. doi: 10.1161/ATVBAHA.109.200873. Epub 2010 Apr 8. PMID 20378849
- [Result] Ji R, Cheng Y, Yue J, Yang J, Liu X, Chen H, Dean DB, Zhang C. MicroRNA expression signature and antisense-mediated depletion reveal an essential role of MicroRNA in vascular neointimal lesion formation. Circ Res. 2007 Jun 8;100(11):1579-88. doi: 10.1161/CIRCRESAHA.106.141986. Epub 2007 May 3. PMID 17478730
- [Result] Sato T, Iwasaki Y, Kikkawa Y, Fukagawa M. An efficacy of intensive vitamin D delivery to neointimal hyperplasia in recurrent vascular access stenosis. J Vasc Access. 2016 Jan-Feb;17(1):72-7. doi: 10.5301/jva.5000469. Epub 2015 Sep 30. PMID 26429127
- [Result] Inoue T, Sata M, Hikichi Y, Sohma R, Fukuda D, Uchida T, Shimizu M, Komoda H, Node K. Mobilization of CD34-positive bone marrow-derived cells after coronary stent implantation: impact on restenosis. Circulation. 2007 Feb 6;115(5):553-61. doi: 10.1161/CIRCULATIONAHA.106.621714. Epub 2007 Jan 29. PMID 17261663
- [Result] Hur J, Yang HM, Yoon CH, Lee CS, Park KW, Kim JH, Kim TY, Kim JY, Kang HJ, Chae IH, Oh BH, Park YB, Kim HS. Identification of a novel role of T cells in postnatal vasculogenesis: characterization of endothelial progenitor cell colonies. Circulation. 2007 Oct 9;116(15):1671-82. doi: 10.1161/CIRCULATIONAHA.107.694778. Epub 2007 Oct 1. PMID 17909106
- [Result] Rodrigues-Diez R, Lavoz C, Carvajal G, Rayego-Mateos S, Rodrigues Diez RR, Ortiz A, Egido J, Mezzano S, Ruiz-Ortega M. Gremlin is a downstream profibrotic mediator of transforming growth factor-beta in cultured renal cells. Nephron Exp Nephrol. 2012;122(1-2):62-74. doi: 10.1159/000346575. Epub 2013 Mar 14. PMID 23548835
- [Result] Maciel TT, Melo RS, Schor N, Campos AH. Gremlin promotes vascular smooth muscle cell proliferation and migration. J Mol Cell Cardiol. 2008 Feb;44(2):370-9. doi: 10.1016/j.yjmcc.2007.10.021. Epub 2007 Nov 12. PMID 18086474
- [Result] Ravelli C, Mitola S, Corsini M, Presta M. Involvement of alphavbeta3 integrin in gremlin-induced angiogenesis. Angiogenesis. 2013 Jan;16(1):235-43. doi: 10.1007/s10456-012-9309-6. Epub 2012 Sep 30. PMID 23053782
- [Derived] Lozano I, Bangueses R, Rodriguez I, Pevida M, Rodriguez-Aguilar R, Rodriguez D, Espasandin-Arias M, Llames S, Meana A, Suarez A, Rodriguez-Carrio J. In-stent restenosis is associated with proliferative skin healing and specific immune and endothelial cell profiles: results from the RACHEL trial. Front Immunol. 2023 May 31;14:1138247. doi: 10.3389/fimmu.2023.1138247. eCollection 2023. PMID 37325628